CLINICAL TRIAL: NCT03119818
Title: Intracellular Phosphate and Adenosine Triphosphate (ATP) Concentration Evolution by Magnetic Resonance (MR) Spectroscopy in Patients During Hemodialysis
Brief Title: Intracellular Phosphate Concentration Evolution During Hemodialysis by MR Spectroscopy
Acronym: CIPHEMO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 69HCL17_0047
Record Dates: First submitted 2017-04-11; First posted 2017-04-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: End-Stage Renal Disease (ESRD)
Keywords: ESRD; hemodialysis; phosphate; ATP; magnetic resonance spectroscopy
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Magnetic Resonance Spectroscopy; Renal Dialysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients suffering from ESRD treated by chronic hemodialysis (Experimental): Patients aged from 18 to 80 years old, suffering from ESRD, treated by chronic hemodialysis since at least 6 months and whose phosphatemia at the beginning of HD sessions ranged from 1.5 to 3 mmol/L. Phosphorus (31P) magnetic resonance spectroscopy will be performed in these patients during hemodialysis in order to measure intracellular phosphate and ATP concentrations and intracellular pH evolution during hemodialysis.
  Interventions: Device: Phosphorus (31P) magnetic resonance spectroscopy; Other: Hemodialysis

INTERVENTIONS:
Device: Phosphorus (31P) magnetic resonance spectroscopy — Phosphorus MR spectroscopy realized using a 3-Tesla MR imaging system. A twenty-cm circular surface coil will be set to the 31P resonance frequency and placed over the leg muscle region to obtain spectroscopy acquisitions. 31P MR spectra will be acquired before, during (every 160 seconds), and 30 minutes after dialysis. 31P MR system data will be analyzed using jMRUI Software. Five different peaks will be analyzed: inorganic phosphate, phosphocreatine, α-, β-, and γ-ATP.
Other: Hemodialysis — Hemodialysis realized using a 5008 generator, a portable plant, a FX80 Dialyzer, a dialyzing solution with a standard electrolytes composition. The dialysis generator will be placed outside of the MRI examination room. The dialysis lines will pass through a wave guide to connect patients positioned on the bed of the MRI. A suitably trained nurse will proceed to the cannulation of the fistula, the connection of the catheter, and the monitoring of the clinical tolerance of the session.

SUMMARY:
End-stage renal disease is associated with hyperphosphatemia due to a decrease of renal phosphate excretion. This hyperphosphatemia is associated with an increase of cardiovascular risk and mortality. Thus, three therapeutic options have been developed: dietary restriction, administration of phosphate binders and phosphorus clearance by hemodialysis (HD).

During a standard HD session, around 600 to 700mg phosphate is removed from the plasma, whereas it contains only 90 mg inorganic phosphate (Pi); 85% of phosphate is stored in bones and teeth in hydroxyapatite form, 14% is stored in the intracellular space (90% organic phosphate and 10% Pi), and 1% remains in the extracellular space.

Currently, the source of Pi cleared during HD remains to be determined. Phosphorus (31P) magnetic resonance spectroscopy allows reliable, dynamic and non-invasive measurements of phosphate intracellular concentration. The investigator's team recently published data obtained in anephric pigs, suggesting that phosphate intracellular concentration increases during a HD session. In parallel, we showed that ATP intracellular concentration decreased. These results suggest that the source of Pi cleared during HD could be located inside the cell.

In this study, investigators will measure intracellular phosphate and ATP concentrations and intracellular potential of hydrogen (pH) evolution during hemodialysis in 12 patients suffering from end-stage renal disease by MR spectroscopy.

If these results were confirmed in humans, it could explain, at least in part, HD intolerance in some patients and would lead to modify therapeutic approaches of hyperphosphatemia, for example, by modifying HD sessions time.

ELIGIBILITY:
Inclusion Criteria:

* Patient suffering from end-stage renal disease, treated by chronic hemodialysis since at less 6 months
* Phosphatemia (at the start of the session) ≥ 1,5 mmol/L and ≤ 3 mmol/L
* written consent signed

Exclusion Criteria:

* Major subject protected by law
* Prisoners or subjects who are involuntarily incarcerated
* Denutrition (weight loss ≥ 5 kg in one months/10 kg in 6 months, Body Mass Index (BMI) ≤ 21 kg/m2, albuminemia ≤ 35 g/L)
* Obesity (BMI ≥ 30 kg/m2)
* Phosphatemia at the start of the dialysis < 1,5 mmol/L or > 3 mmol/L
* Secondary hyperparathyroidism with parathormone (PTH) ≥ 1000 pg/mL
* Adynamic osteopathy (PTH ≤ 50 pg/mL)
* Hypoparathyroidism with a history of parathyroidectomy
* Hemoglobin ≤ 100 g/L
* Contraindication to heparin
* Temporary vascular access
* Contraindication to resonance magnetic spectroscopy (pacemaker or insulin pump, metallic valvular prosthesis, valvular prosthesis not compatible with resonance magnetic spectroscopy, dental appliance, intracerebral clip, claustrophobic subject).
* Simultaneous participation to another research protocol
* Patient not affiliated to a social security system

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2017-06-14 (Actual); Primary Completion 2017-07-29 (Actual); Study Completion 2017-07-29 (Actual)

PRIMARY OUTCOMES:
Change in phosphate intracellular concentration | Baseline, at start of HD, every 160 seconds during HD, at the end of HD and 30 minutes after HD
  Measurement of phosphate intracellular concentration evolution during a 4 hours hemodialysis (HD) session using phosphorus magnetic resonance spectroscopy.

SECONDARY OUTCOMES:
Change in ATP intracellular concentration | Baseline, at start of HD, every 160 seconds during HD, at the end of HD and 30 minutes after HD
  Measurement of ATP intracellular concentration evolution during a 4 hours HD session using phosphorus magnetic resonance spectroscopy.
Change in intracellular pH | Baseline, at start of HD, every 160 seconds during HD, at the end of HD and 30 minutes after HD
  Measurement of intracellular pH evolution during a 4 hours HD session using phosphorus magnetic resonance spectroscopy. Intracellular pH will be calculated using the Henderson-Hasselbach formula: Ph = 6.75 + log (δ-3.27)/(5.69-δ), with δ being the difference (in parts per million) between inorganic phosphate (Pi) and phosphocreatine (PCr) resonance frequencies.
Change in phosphatemia | At start of HD, every 15 minutes during first hour of HD, then every hour during HD, at the end of HD and 30 minutes after HD
  Measurement of intracellular pH evolution during a 4 hours HD session using phosphorus magnetic resonance spectroscopy. Intracellular pH will be calculated using the Henderson-Hasselbach formula: Ph = 6.75 + log (δ-3.27)/(5.69-δ), with δ being the difference (in parts per million) between Pi (inorganic phosphate) and PCr (phosphocreatine) resonance frequencies.
Calcium balance | At the end of a 4 hours HD session
  Calcium balance will be measured using the formula: (Cae - Cab)(Ve - UF)+(Cae * UF), where Cae is the calcium in the efﬂuent, Cab is the calcium in the dialysis solution, Ve is the volume of efﬂuent, and UF is the ultraﬁltration.

CONTACTS AND LOCATIONS:
Overall Officials: Laurent JUILLARD, MD, PhD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Service de Néphrologie Pavillon P, Hôpital E. Herriot, Lyon, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chazot G, Lemoine S, Kocevar G, Kalbacher E, Sappey-Marinier D, Rouviere O, Juillard L. Intracellular Phosphate and ATP Depletion Measured by Magnetic Resonance Spectroscopy in Patients Receiving Maintenance Hemodialysis. J Am Soc Nephrol. 2021 Jan;32(1):229-237. doi: 10.1681/ASN.2020050716. Epub 2020 Oct 22. PMID 33093193